CLINICAL TRIAL: NCT04590027
Title: Caudal Block Versus Local Wound Infiltration for Inguinal Procedures in Young Children. A Prospective Observational Trial
Brief Title: Caudal Block Versus Local Wound Infiltration for Inguinal Procedures
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: 621/2013BO1
Record Dates: First submitted 2020-09-16; First posted 2020-10-19 (Actual); Results first posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2020-08

CONDITIONS: Anesthesia, Caudal
Keywords: caudal block; wound infiltration; postoperative pain; outpatient surgery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Single-centre observational study to analyse whether there is a difference in post-operative pain scores and set up time when comparing caudal block with local wound infiltration

DETAILED DESCRIPTION:
Inguinal procedures in children are surgical frequently performed in an outpatient setting. This study analyzed regional analgesia for inguinal procedures in toddlers comparing caudal block with local wound infiltration and assessed post-operative pain scores as well as process times.A number of documents were compiled to inform and record data: a standard anaesthesia protocol, a documentation sheet for intraoperative recording, an information leaflet for the parents and a documentation sheet for the post-operative course of 24 hours .

Caudal anaesthesia was performed after induction of anaesthesia. In patients getting wound infiltration ropivacaine 0.375% 0.5 ml kg-1 was injected subcutaneously after closing of the fascia transversalis.

Parents were informed about the study and invited to participate upon arriving on the outpatient ward if the patient fulfilled the following inclusion criteria: scheduled for elective inguinal procedure, age three to 72 months, no contraindication for either local or caudal analgesia, no comorbidities. If parents agreed to participate, written informed consent was obtained. Pain score and administration of analgesics, vomiting, interval until micturition and interval until mobilization as well as sleep quality during the first post-operative night were documented by the parents in the provided booklet.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* no return of questionnaire
* parents do not understand language

Ages: 3 Months to 68 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: outpatient setting
  paediatric inguinal procedures classifeind ASA 1 or 2 perfomed from the department of paediatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2014-02-01 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2020-01-30 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The clinical trial was conducted at the University Hospital of Tuebingen, Germany, where paediatric inguinal procedures in children classified as ASA I or ASA II ( American Society of Anesthesiologists Physical Status System) are performed in an outpatient setting. Recruitment period:Between February 2014 and June 2015,
Pre-assignment Details: Causes for exclusion from the study No return of Questionaire (n=31) Not meeting criteria for anaesthesia (n=3)
Groups:
- Caudal Block: Caudal anaesthesia was performed after induction of anaesthesia. The puncture site was preoperatively anesthetized with Eutetic Mixture of Local Anaesthetics (EMLA®). The patient was then placed in a lateral decubitus position with left side down. An Epican® Paed 23G Tuohy needle was inserted into the epidural space using anatomical landmarks. After negative aspiration, a combination of a local anaesthetic (1 ml kg-1 ropivacaine 0,2%) and clonidine (2 μg kg-1) was applied.
- Local Infiltration (LI): In patients randomised to the Local Infiltration group (LI) ropivacaine 0.375% 0.5 ml kg-1 was injected subcutaneously after closing of the fascia transversalis.
Period: Overall Study
Arm/Group | Caudal Block | Local Infiltration (LI)
Started | 47 | 39
Completed | 30 | 22
Not Completed | 17 | 17
Not completed — Lost to Follow-up | 17 | 14
Not completed — Protocol Violation | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Caudal Block (CB): Caudal Block (CB)
  pain management
  1 ml kg-1 ropivacaine and clonidine 2 ug kg-1
- Local Infiltration (LI): Local Infiltration (LI) pain management 0.375% 0.5 ml kg-1 ropivacaine injected subcutaneously
- Total: Total of all reporting groups
Arm/Group | Caudal Block (CB) | Local Infiltration (LI) | Total
Number analyzed (Participants) | 47 | 39 | 86
Age, Continuous [Mean (Standard Deviation); unit: month] — Population: The random sample was 52 patients. 34 patients were excluded.
  month
    number analyzed (Participants) | 30 | 22 | 52
    (all) | 21 (14.7) | 30 (18.8) | 25.5 (16.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 44 | 35 | 79
Region of Enrollment [Number; unit: participants]
  Germany | 47 | 39 | 86
Weight of Children [Median (Inter-Quartile Range); unit: kilogram] — weight measured in kg Population: Thirty-one patients had to be excluded from the analysis because the parents did not return the questionnaire. Another three patients were excluded because the specified anaesthesia protocol was not followed.
  kilogram
    number analyzed (Participants) | 30 | 22 | 52
    (all) | 10 [6.5 to 18] | 12 [8.2 to 24] | 11 [6.5 to 24]

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Analgesia Quality Between the Two Groups
Description: Visual Analog Score (VAS) Minimum 0 (no pain) and Maximum 10 (worst pain) A two point difference of mean pain scores was defined as clinically meaningful to establish a superiority for one of the procedures of pain management
Time Frame: Arrival on postoperative care unit (PCU), arrival ward, 1h, 2 h 3h, 4h, 5h, 6h, 12h. 24h,
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Caudal Block: Ropivacaine 0,2 % 1 ml kg-1 and clonidine 2 μg kg-1
- Local Infiltration: Ropivacaine 0.375% 0.5 ml kg-1 was injected subcutaneously
Arm/Group | Caudal Block | Local Infiltration
Number analyzed (Participants) | 30 | 22
score on a scale
  Arrival PCU | 1.86 (0.43) | 3.09 (0.51)
  Arrival ward | 1.83 (0.5) | 2.95 (0.58)
  1h | 1.36 (0.31) | 2.13 (0.37)
  2h | 1.3 (0.33) | 1.68 (0.39)
  3h | 1.43 (0.31) | 1.54 (0.36)
  4h | 2.0 (0.34) | 0.86 (0.40)
  5h | 1.76 (0.34) | 0.77 (0.40)
  6h | 1.5 (0.28) | 1.00 (0.33)
  12h | 1.56 (0.35) | 1.31 (0.41)
  24 h | 0.56 (0.22) | 0.68 (0.26)
Statistical Analysis 1: Comparison: Caudal Block vs Local Infiltration; Test type: Non-Inferiority — power calculation was not recorded Definition of non inferiority: two point difference of pain score at the measurement times; p < 0.05, ANCOVA; To rule out confounders due to an age difference, the ANCOVA test was applied to compare the differences in pain scores age-unrelatedly; Fisher Yates Test to compare the requirement of resue medication

2. Secondary Outcome: Set up Time
Description: How much times goes by for induction of anesthesia in both groups
Time Frame: Time in minutes measured between start of induction of anesthesia to start of surgical incision
Population: to analyze which procedure is less time consuming
Measure: Median (Inter-Quartile Range); unit: minutes
Groups:
- Caudal Block: Ropivacaine 0,2% 1ml kg-1 and clonidine 2µg kg-1
- Local Infiltration: Ropivacaine 0.375% 0.5 ml kg-1 subcutaneously
Arm/Group | Caudal Block | Local Infiltration
Number analyzed (Participants) | 30 | 22
minutes | 22.5 [16 to 46] | 17 [10 to 35]
Statistical Analysis 1: Comparison: Caudal Block vs Local Infiltration; Test type: Superiority; p < 0.05, Chi-squared

3. Secondary Outcome: Rescue Medication
Description: total number of analgesic doses across all participants
Time Frame: 24 hours
Population: The need for rescue medicine is an indirect parameter for the effectiveness of the analgesic procedure.
Measure: Number; unit: total number analgesic dosis
Groups:
- Caudal Block: ropivacaine 0,2% 1 ml kg-1 and clonidine 2 μg kg-1
- Local Infiltration: Ropivacaine 0.375% 0.5 ml kg-1
Arm/Group | Caudal Block | Local Infiltration
Number analyzed (Participants) | 30 | 22
total number analgesic dosis | 58 | 31

4. Secondary Outcome: Neurological Outcome
Description: Time until first micturation an time to motor activity
Time Frame: 24 hours
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 0-24 h postoperatively
Groups:
- Caudal Block: Caudal anaesthesia was performed after induction of anaesthesia. The puncture site was preoperatively anesthetized with EMLA®. The patient was then placed in a lateral decubitus position with left side down. An Epican® Paed 23G Tuohy needle was inserted into the epidural space using anatomical landmarks. After negative aspiration, a combination of a local anaesthetic (1 ml kg-1 ropivacaine 0,2%) and clonidine (2 μg kg-1) was applied.
- Local Infiltration: In patients randomised to the LI group ropivacaine 0.375% 0.5 ml kg-1 was injected subcutaneously after closing of the fascia transversalis.
Arm/Group | Caudal Block | Local Infiltration
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/22
Other Adverse Events (participants affected / at risk) | 2/30 | 3/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caudal Block (N=30) | Local Infiltration (N=22)
vomiting (Gastrointestinal disorders) | 2 (2) | 3 (3) — vomiting
delayed micturation (Renal and urinary disorders) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Since postoperative pain and emergence delirium might overlap within the first half hour after the procedure, a paediatric anaesthesia emergence delirium scale might have been useful.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No